CLINICAL TRIAL: NCT00407667
Title: Transcranial Direct Current Stimulation (tDCS) of the Lesioned or Non-lesioned Hemisphere Plus Computer-assisted Arm Trainer: a Randomized, Placebo-controlled Double-blind Multi-centre Study in Patients With Severe Arm Paresis Early After Stroke
Brief Title: Transcranial Galvanic Stimulation After Stroke
Acronym: TraGAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: TraGAT, Charité - University Medicine Berlin
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TraGAT
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2006-11

CONDITIONS: Stroke
Keywords: hemiparesis; rehabilitation; upper limb rehabilitation; arm therapy
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): patients receive 20 min of anodal transcranial stimulation plus 20 min of repetitive arm training with a therapy robot(Bi-Manu-Track)
  Interventions: Device: transcranial galvanic stimulation
- 2 (Experimental): patients receive 20 min of cathodal transcranial stimulation plus 20 min of repetitive arm training with a therapy robot(Bi-Manu-Track)
  Interventions: Device: transcranial galvanic stimulation
- 3 (Sham Comparator): patients receive 20 min of sham transcranial stimulation plus 20 min of repetitive arm training with a therapy robot(Bi-Manu-Track)
  Interventions: Device: transcranial galvanic stimulation

INTERVENTIONS:
Device: transcranial galvanic stimulation — for tDCS: Siemens Universal-Neuroton 826 for arm training: Bi-Manu-Track, Reha-Stim, Berlin

SUMMARY:
Transcranial galvanic stimulation (tDCS) seems to promote motor recovery after stroke by stimulating (anodal) or inhibiting (cathodal) neural circuits in the brain. In the treatment of severe arm paresis after stroke, robot-assisted arm training (AT) proved to be effective, but nevertheless only a few patients could use their affected hand functionally in daily life after robot training. Therefore the present study intends to combine both approaches, tDCS + AT, applied at the same time every day for six weeks. The study has three treatment arms, two groups will receive the tDCS, either anodal of the lesioned or cathodal of the non-lesioned hemisphere. The anodal stimulation is expected to facilitate the activity of the arm motor area of the lesioned side directly, while the cathodal stimulation of the non-lesioned hemisphere is expected to facilitate the lesioned side indirectly by decreasing inhibitory inputs. The third group will receive a sham-stimulation. All patients will work with the AT simultaneously to the tDCS, respectively sham-tDCS.

ELIGIBILITY:
Inclusion Criteria:

* subacute stroke
* stroke interval 3 to 8 weeks
* severe upper limb paresis
* Fugl-Meyer < 18

Exclusion Criteria:

* history of epilepsy
* antiepileptic, neuroleptic medication
* metal implants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Limb Motor Score (0-66) | 45 min

SECONDARY OUTCOMES:
Box&Block Test | 5 min

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hesse, MD, Principal Investigator — Charité -University Medicine Berlin; Medical Park Berlin
Locations (3):
- Germany (2):
  - Charité, University Medicine Berlin, Medical Park Berlin, Berlin
  - Klinik Bavaria, Kreischa
- Villa Melitta, Bolzano, Italy